CLINICAL TRIAL: NCT02482155
Title: Pharmacokinetic Study of a Single Oral Administration of MOMENT ACT ANALGESIC Granules for Oral Solution to Healthy Volunteers Under Fasting Conditions Single Centre, Single Dose, Open-label, Bioavailability Study
Brief Title: Ibuprofen (MOMENT ACT ANALGESIC Granules) Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 070(I)HO14386; CRO-PK-14-291 (Other: CROSS Research S.A., Phase I Unit)
Record Dates: First submitted 2015-06-17; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: pharmacokinetics; MOMENTACT; ibuprofen 400 mg; oral; granules
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ibuprofen (Experimental): ibuprofen 400 mg granules, oral solution, single administration under fasting conditions
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — ibuprofen 400 mg single dose oral solution
  Other Names: MOMENTACT

SUMMARY:
The main purpose of this study was to evaluate the pharmacokinetic (PK) profile of ibuprofen after oral administration of a single dose of MOMENT ACT ANALGESIC granules to healthy male and female subjects, under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study;
2. Sex and age: females and males, 18-55 years old both inclusive;
3. Body Mass Index (BMI): 18.5-30 kg/m2 inclusive;
4. Vital signs: systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, heart rate (HR) 50-90 bpm, measured after 5 min at rest in the sitting position;
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study;
6. Contraception and fertility (females only): females of child-bearing potential must be using at least one of the following reliable methods of contraception:

   1. hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit;
   2. a non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit;
   3. a male sexual partner who agrees to use a male condom with spermicide;
   4. a sterile sexual partner. Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all female subjects, pregnancy test result must be negative at screening and day -1.

Exclusion Criteria:

1. Electrocardiogram (ECG) 12-leads (supine position): clinically significant abnormalities;
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study;
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness;
4. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients or related drugs, namely non-steroidal anti-inflammatory agents (NSAIDs); history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study;
5. Diseases: history of significant renal, hepatic, gastrointestinal (in particular gastroduodenal ulcer and bleeding), cardiovascular, respiratory (in particular asthma), skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study;
6. Medications: medications, including over the counter (OTC) medications and herbal products for 2 weeks before the start of the study, in particular ibuprofen. Hormonal contraceptives for females are allowed;
7. Investigative drug studies: participation in the evaluation of any investigational product in the 3 months before this study, calculated from the first day of the month following the last visit of the previous study;
8. Blood donation: blood donations in the 3 months before this study;
9. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to United States Department of Agriculture Dietary Guidelines 2010], caffeine (>5 cups coffee/tea/day) or tobacco abuse (>=10 cigarettes/day); daily use of distilled spirits;
10. Drug test: positive result at the drug test at screening or day-1;
11. Alcohol test: positive alcohol breath test at day -1;
12. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study, vegetarians;
13. Pregnancy (females only): positive or missing pregnancy test at screening or day -1, pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of ibuprofen | 0, 3, 5, 10, 15, 20, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24 hours post-dose
Area under the plasma concentration versus time curve (AUC) of ibuprofen | 0, 3, 5, 10, 15, 20, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24 hours post-dose
Time to Cmax (Tmax) of ibuprofen | 0, 3, 5, 10, 15, 20, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24 hours post-dose
Apparent terminal elimination rate constant (λz) of ibuprofen | 0, 3, 5, 10, 15, 20, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24 hours post-dose
Apparent terminal elimination half-life (t1/2,z) of ibuprofen | 0, 3, 5, 10, 15, 20, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24 hours post-dose
Lag-time from the dosing time point prior to the first measurable plasma concentration (tlag) of ibuprofen | 0, 3, 5, 10, 15, 20, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24 hours post-dose
Time to the first ibuprofen plasma concentration of 5 ug/mL (ton5) | 0, 3, 5, 10, 15, 20, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24 hours post-dose

SECONDARY OUTCOMES:
Time to the first ibuprofen plasma concentration of 10 ug/mL (ton10) | 0, 3, 5, 10, 15, 20, 30, 45 minutes, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, 24 hours post-dose
Occurrence of adverse effects | up to 24 hours after administration

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — Cross Research S.A.
Locations (1):
- CROSS Research S.A., Phase I Unit, Via F.A. Giorgioli 14 Phone: Fax: +41.91.63.00.511 Email:, Arzo, Switzerland